CLINICAL TRIAL: NCT04128475
Title: Long-term Study of LDL-c Lowering With Evolocumab: Observational Follow-up After the FOURIER OUTCOMES Trial.
Brief Title: Observational Study of Cardiovascular Disease.
Acronym: FOURIER LEGACY
Status: Terminated | Type: Observational
Why Stopped: Withdrawal of funding.
Sponsor: University of Sydney (Other)
Collaborators: The TIMI Study Group (Other); Imperial College London (Other); University of Oslo (Other); Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CTC0173
Record Dates: First submitted 2019-09-12; First posted 2019-10-16 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Cardiovascular Morbidity; Coronary Heart Disease; Low-density-lipoprotein-type
Keywords: Cardiovascular events; Coronary heart disease; Cardiovascular death; Low density lipoprotein cholesterol (LDL-c); Evolocumab; FOURIER OUTCOMES
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: N/A - observational study. — N/A - observational study.

SUMMARY:
This observational study will follow participants who completed follow-up in the FOURIER OUTCOMES trial to evaluate the long-term effects of evolocumab treatment. Long-term post-trial (legacy) beneficial effects have been reported with statins, niacin, hypoglycemic therapy and fibrates. Whether similar effects are seen after LDL cholesterol (LDL-c) lowering by PCSK9 inhibition is currently unknown.

Evolocumab therapy causes a profound reduction in LDL cholesterol of approximately 60%. Statins have shown legacy effects over 5 years post-trial, including a 7% reduction in total mortality in meta-analysis and 12% reduction in coronary mortality. It would therefore be hypothesized that additional effects beyond the trial period would be conferred by previous evolocumab treatment. It is also important to assess the long-term safety of prior evolocumab treatment.

ELIGIBILITY:
Subjects who completed the FOURIER OUTCOMES trial (defined as attendance at close-out visit irrespective of treatment compliance) will be approached by FOURIER OUTCOMES site investigators and asked about their interest in taking part in this trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in selected countries who completed the FOURIER OUTCOMES trial, irrespective of non-fatal on-study events during FOURIER OUTCOMES trial, and who agree to take part in the FOURIER LEGACY study following study completion will be enrolled into this trial.
Sampling Method: Non-Probability Sample
Enrollment: 1137 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
To evaluate the potential long-term effect of evolocumab treatment on a composite of CV death, MI, stroke or coronary revascularisation in participants completing participation in the FOURIER OUTCOMES trial. | 5 years
  To evaluate the potential long-term effect of evolocumab treatment on a composite of CV death, MI, stroke or coronary revascularization in patients completing participation in the FOURIER OUTCOMES trial.

SECONDARY OUTCOMES:
To evaluate the potential long-term effect of evolocumab treatment on a composite of CV death, MI, stroke or coronary revascularization in patients completing participation in the FOURIER OUTCOMES trial. | 5 years
  To evaluate the potential long-term effect of evolocumab treatment on a composite of CV death, MI, stroke or coronary revascularization in patients completing participation in the FOURIER OUTCOMES trial.
To evaluate the long-term effect of evolocumab treatment on CV death. | 5 years
  To evaluate the long-term effect of evolocumab treatment on CV death.
To evaluate the long-term effects of evolocumab treatment on CHD death. | 5 years
  To evaluate the long-term effects of evolocumab treatment on CHD death.
To evaluate the long-term effect of evolocumab treatment on the individual components of the primary endpoint and any other CV hospitalizations. | 5 years
  To evaluate the long-term effect of evolocumab treatment on the individual components of the primary endpoint and any other CV hospitalizations.
To evaluate the long-term effect of evolocumab treatment on amputations and peripheral revascularization. | 5 years
  To evaluate the long-term effect of evolocumab treatment on amputations and peripheral revascularization.
To evaluate the long-term effect of evolocumab treatment in terms of all-cause death (and non-CV, including cancer, death). | 5 years
  To evaluate the long-term effect of evolocumab treatment in terms of all-cause death (and non-CV, including cancer, death).
To assess the effect modification of use or prescription lipid-lowering treatment classes (statins, cholesterol absorption inhibitors, PCSK9i) administered at FOURIER OUTCOMES trial entry on the outcomes above. | 5 years
  To assess the effect modification of use or prescription lipid-lowering treatment classes (statins, cholesterol absorption inhibitors, PCSK9i) administered at FOURIER OUTCOMES trial entry on the outcomes above.
To assess the effect modification by baseline characteristics on defined study outcomes above. | 5 years
  To assess the effect modification by baseline characteristics on defined study outcomes above.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Keech, Study Chair — National Health and Medical Research Council, Australia; Peter Sever, Study Chair — Imperial College London
Locations (3):
- TIMI Study Group, Boston, Massachusetts, United States
- Oslo University Hospital, Nydalen, Oslo County, Norway
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No